CLINICAL TRIAL: NCT01054170
Title: A 12-week, Phase II, Double-blind, Placebo-Controlled, Randomised, Parallel-Group, Multi-Centre Study to Assess the Effect of 60mg AZD9668 Administered Orally Twice Daily on Structural Changes in the Airways by Multi-Slice Computed Tomography in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Effect on Structural Changes in Airways, Measured by MSCT, of Twice Daily 60mg AZD9668 for 12 Weeks in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0520C00014
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2012-07-25 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic; obstructive; pulmonary; lung; respiratory disease; efficacy; placebo-controlled; COPD; FEV1; St Georges Respiratory Questionnaire; Computed Tomography; MSCT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Respiration Disorders | interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD9668 (Experimental)
  Interventions: Drug: AZD9668
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9668 — 2 x 30 mg oral tablets twice daily (bid) for 12 weeks
  Arms: AZD9668
Drug: Placebo — 2 x matched placebo to oral tablet twice daily (bid) for 12 weeks
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate structural changes effected by AD9668 in the airways of adults with Chronic Obstructive Pulmonary Disease (COPD) by Multi-Slice Computed Tomography (MSCT)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD with symptoms over 1 year
* FEV1/FVC < 70% and FEV1 >= 40 and < =70 % of predicted post-bronchodilator
* Ex-smokers for at least 12 months

Exclusion Criteria:

* Past history or current evidence of clinically significant heart disease
* Current diagnosis of asthma
* Worsening of COPD requiring hospitalisation and/or treatment with antibiotics and/or an increase in inhaled steroid dose and/or oral steroids within 4 weeks of study visit 1b

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Asger Dirksen, Principal Investigator — Gentofte Hospital, Department of Lung Medicine
Locations (9):
- Canada (2):
  - Research Site, Kingston, Ontario
  - Research Site, Québec, Quebec
- Denmark (3):
  - Research Site, Hellerup
  - Research Site, Hvidovre
  - Research Site, Odensec
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Nieuwegein
- Research Site, Bucharest, Romania
- Research Site, Kyiv, Ukraine

REFERENCES:
- [Derived] Nordenmark LH, Taylor R, Jorup C. Feasibility of Computed Tomography in a Multicenter COPD Trial: A Study of the Effect of AZD9668 on Structural Airway Changes. Adv Ther. 2015 Jun;32(6):548-66. doi: 10.1007/s12325-015-0215-3. Epub 2015 Jun 5. PMID 26043724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 06 January 2010; Last patient completed: 17 November 2010; Twelve centres across 5 countries participated in this study: Canada (2), Denmark (3), The Netherlands (2), Romania (2) and Ukraine (3).
Pre-assignment Details: Tiotropium maintenance therapy and reliever medication were commenced at screening, except for patients on inhaled corticosteroids (ICS, ICS/LABA) who were required to stop these at enrolment and commence on tiotropium and reliever medication at the same time. These patients received tiotropium for a period of at least 3 weeks before screening.
Groups:
- AZD9668: AZD9668 2x30mg bid
- Placebo: Placebo 2 tablets bid
Period: Overall Study
Arm/Group | AZD9668 | Placebo
Started | 25 | 27
Completed | 21 | 21
Not Completed | 4 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9668 | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age Continuous [Mean (Standard Deviation); unit: years] | 7.2 (65) | 7.7 (66) | 7.45 (131)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: AWT-Pi10 (Airway Wall Thickness of a Theoretical Airway With an Internal Perimeter of 10 mm)
Description: AWT-Pi10 (mm) as a measure of structural changes in airways. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: The efficacy analysis set for each outcome measure includes those patients who received at least one dose of investigational product and for whom a baseline and at least one post-randomisation measurement is available for that outcome measure. Patients were analysed by to randomised treatment in accordance with the intention to treat principle.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 17 | 19
mm | 3.84 (0.021) [lower limit 0.021] | 3.83 (0.017) [lower limit 0.017]

2. Secondary Outcome: 5th Generation Wall Area Percentage
Description: 5th Generation Wall Area Percentage as a measure of structural changes in airways. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage Area
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 17 | 19
Percentage Area | 66.21 (0.275) [lower limit 0.275] | 65.94 (0.234) [lower limit 0.234]

3. Secondary Outcome: Air Trapping Index (ATI) on Expiratory Scans
Description: ATI Percentage as a measure of structural changes in airways. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ATI Percentage
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 15 | 13
ATI Percentage | 54.56 (1.706) [lower limit 1.706] | 57.12 (1.599) [lower limit 1.599]

4. Secondary Outcome: Pre-bronchodilator Inspiratory Capacity (IC)
Description: Inspiratory Capacity (L) as a measure of lung function. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 23
L | 2.56 (0.154) [lower limit 0.154] | 2.39 (0.153) [lower limit 0.153]

5. Secondary Outcome: Pre-bronchodilator Total Lung Capacity (TLC)
Description: Total Lung Capacity (L) as a measure of lung function. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 23
L | 7.03 (0.178) [lower limit 0.178] | 6.92 (0.177) [lower limit 0.177]

6. Secondary Outcome: Pre-bronchodilator Functional Residual Capacity (FRC)
Description: Functional Residual Capacity (L) as a measure of lung function. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 23 | 23
L | 4.41 (0.165) [lower limit 0.165] | 4.21 (0.158) [lower limit 0.158]

7. Secondary Outcome: Pre-bronchodilator Residual Volume (RV)
Description: Residual volume (L) as a measure of lung function. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 23
L | 3.64 (0.161) [lower limit 0.161] | 3.73 (0.161) [lower limit 0.161]

8. Secondary Outcome: Pre-bronchodilator Specific Airway Conductance (SGaw)
Description: Specific Airway Conductance as a measure of lung function. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: 1/[s*kPa]
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 23
1/[s*kPa] | 0.52 (0.034) [lower limit 0.034] | 0.48 (0.034) [lower limit 0.034]

9. Secondary Outcome: Pre-bronchodilator Diffusion Capacity of Carbon Monoxide (DLco)
Description: Capacity of Carbon Monoxide as a measure of lung function. End of treatment Least Squares Mean.
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/kPa*min
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 23 | 23
mmol/kPa*min | 5.49 (0.204) [lower limit 0.204] | 5.67 (0.209) [lower limit 0.209]

10. Secondary Outcome: Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic. End of treatment value or Last Observation Carried Forward (LOCF).
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
L | 1.51 (0.048) [lower limit 0.048] | 1.49 (0.050) [lower limit 0.050]

11. Secondary Outcome: Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic. End of treatment value or Last Observation Carried Forward (LOCF).
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 21 | 23
L | 1.60 (0.050) [lower limit 0.050] | 1.58 (0.050) [lower limit 0.050]

12. Secondary Outcome: Pre-bronchodilator Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (L) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic. End of treatment value or Last Observation Carried Forward (LOCF).
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
L | 3.25 (0.084) [lower limit 0.084] | 3.14 (0.083) [lower limit 0.083]

13. Secondary Outcome: Post-bronchodilator Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (L) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic. End of treatment value or Last Observation Carried Forward (LOCF).
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 21 | 23
L | 3.34 (0.083) [lower limit 0.083] | 3.34 (0.080) [lower limit 0.080]

14. Secondary Outcome: Pre-bronchodilator Slow Vital Capacity (SVC)
Description: Slow Vital Capacity (L) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic. End of treatment value or Last Observation Carried Forward (LOCF).
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
L | 3.42 (0.069) [lower limit 0.069] | 3.38 (0.068) [lower limit 0.068]

15. Secondary Outcome: Post-bronchodilator Slow Vital Capacity (SVC)
Description: Slow Vital capacity (L) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic. End of treatment value or Last Observation Carried Forward (LOCF).
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 21 | 23
L | 3.56 (0.063) [lower limit 0.063] | 3.44 (0.061) [lower limit 0.061]

16. Secondary Outcome: Peak Expiratory Flow (PEF) Morning (Daily Recordings)
Description: Peak Expiratory Flow (L/min) as a measure of lung function, measured at home by the patient each morning.
Time Frame: Average from measurements recorded daily by patient in last 6 weeks of treatment.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
L/min | 255.82 (9.956) [lower limit 9.956] | 244.16 (9.871) [lower limit 9.871]

17. Secondary Outcome: Peak Expiratory Flow (PEF) Evening (Daily Recordings)
Description: Peak Expiratory Flow (L/min) as a measure of lung function, measured at home by the patient each evening .
Time Frame: Average from measurements recorded daily by patient in last 6 weeks of treatment.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
L/min | 264.15 (10.02) [lower limit 10.02] | 254.31 (9.966) [lower limit 9.966]

18. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Morning (Daily Recordings)
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function, measured at home by the patient each morning.
Time Frame: Average from measurements recorded daily by patient in last 6 weeks of treatment.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
L | 1.49 (0.065) [lower limit 0.065] | 1.29 (0.066) [lower limit 0.066]

19. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Evening (Daily Recordings)
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function, measured at home by the patient each evening.
Time Frame: Average from measurements recorded daily by patient in last 6 weeks of treatment.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
L | 1.51 (0.062) [lower limit 0.062] | 1.30 (0.064) [lower limit 0.064]

20. Secondary Outcome: Breathlessness, Cough and Sputum Scale (BCSS) Total Score
Description: Breathlessness, Cough and Sputum Scale, patient reported questionnaire as a measure of respiratory symptoms (reported on a 0 (best health status) to 12 (worst possible status) scale).
Time Frame: Average from measurements recorded daily by patient in last 6 weeks of treatment.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Total Score
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
Total Score | 2.33 (0.319) [lower limit 0.319] | 3.36 (0.301) [lower limit 0.301]

21. Secondary Outcome: EXAcerbations of Chronic Pulmonary Disease Tool (EXACT) Total Score
Description: EXAcerbations of Chronic pulmonary disease Tool, patient questionnaire as a measure of respiratory symptoms (reported as units on a 0 (best health status) to 100 (worst possible status) scale).
Time Frame: Average from measurements recorded daily by patient in last 6 weeks of treatment.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Total Score
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 26
Total Score | 28.48 (2.065) [lower limit 2.065] | 33.26 (2.013) [lower limit 2.013]

22. Secondary Outcome: St George's Respiratory Questionnaire for COPD Patients (SGRQ-C) Overall Score
Description: St George's Respiratory Questionnaire for Chronic Obstructive Pulmonary Disease, as a measure of Quality of Life (reported on a % scale from 0 (best health status) to 100(worst possible status)).
Time Frame: Measured after 12 weeks treatment (day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 23
Scores on a scale | 35.64 (2.364) [lower limit 2.364] | 39.61 (2.389) [lower limit 2.389]

23. Secondary Outcome: Percentage of Reliever Free Days in Last Six Weeks of Treatment
Description: Percentage of reliever free days in last 6 weeks on treatment.
Time Frame: Average from measurements recorded daily by patient in last 6 weeks of treatment.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
percentage of days | 34.23 (6.394) [lower limit 6.394] | 26.43 (6.001) [lower limit 6.001]

24. Secondary Outcome: Exacerbations
Description: Number of patients experiencing disease exacerbations on treatment.
Time Frame: Exacerbations were recorded at all study visits (after 1, 4, 8, and 12 weeks of treatment and at follow up)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 25 | 27
Participants | 0 | 5

ADVERSE EVENTS:
Arm/Group | AZD9668 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/27
Other Adverse Events (participants affected / at risk) | 8/25 | 8/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9668 (N=25) | Placebo (N=27)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9668 (N=25) | Placebo (N=27)
DRY MOUTH (Gastrointestinal disorders) | 0 | 2
ASTHENIA (General disorders) | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 5 | 2
DIZZINESS (Nervous system disorders) | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 3
BRONCHIAL WALL THICKENING (Respiratory, thoracic and mediastinal disorders) | 1 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No